CLINICAL TRIAL: NCT02551939
Title: Magnetic Resonance Imaging and Breast-Q Evaluation After Breast Autologous Fat Grafting Augmentation in Chinese Women
Brief Title: Breast Fat Grafting Augmentation in Chinese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jun Li, Doctor， head of the Department of Plastic & Cosmetic Surgery, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 201352
Record Dates: First submitted 2015-09-13; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Breast Implantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fat graft (Experimental): Autologous Fat Grafting
  Interventions: Procedure: Autologous Fat Grafting

INTERVENTIONS:
Procedure: Autologous Fat Grafting — Autologous Fat Grafting

SUMMARY:
A total of 38 Chinese healthy women underwent autologous fat grafting for cosmetic breast augmentation. Breast volumes were measured by magnetic resonance imaging preoperatively and 1 year after the procedure. Furthermore, BREAST-Q was used to analyze the satisfaction and well-being of patients during the preoperative and 1 year post operation.

DETAILED DESCRIPTION:
Autologous fat was obtained from thighs, waist or abdomen using resonance liposuction instrument. Fat was injected into the tissues in a multitunnel and multilayer way until they were firm and appeared fully tumesced according to the Coleman method.All MRI volume analyses were blindly performed by examiner independently preoperatively and 1 year postoperatively. Object marking was done using avanto 1.5T superconducting magnetic resonance scanner.Volume analysis was done by counting pixels within the frames of the MRI using ImageChecker CAD software.The Chinese version of BREAST-Q augmentation module was obtained from the Memorial Sloan-Kettering Cancer Center and the University of British Columbia. 38 patients were given the BREAST-Q questionnaire to express their thoughts preoperatively and 1 year postoperatively. Data were calculated using the Q-score program, which converts raw BREAST-Q scores of 1 through 4 or 5 to scores of 0 to 100.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women agreed to participate in the study

Exclusion Criteria:

* Patients who had breast surgery previously
* Women on the lactation or gestation period

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Breast volumes were measured by magnetic resonance imaging | one year
BREAST-Questionaire was used to analyze the satisfaction and well-being of patients | one year